CLINICAL TRIAL: NCT07212101
Title: Assessing and Optimizing Sleep, Diet, and Performance in Columbia University Baseball Players
Brief Title: Sleep in Collegiate Baseball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Arizona (Other); Idorsia Pharmaceuticals Ltd. (Industry); Oura Ring (Unknown)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Professor of Nutritional Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAV4501
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Sleep
MeSH Terms: interventions — Sleep; Diet

STUDY DESIGN:
Intervention Model Description: Single group intervention evaluating outcomes pre and post intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep & diet intervention (Experimental): Participants will be asked to increase their fruit and vegetable consumption, time in bed, and modify light exposure across the day
  Interventions: Behavioral: Sleep and diet

INTERVENTIONS:
Behavioral: Sleep and diet — Participants will be asked to increase their fruit and vegetable consumption, time in bed, and modify light exposure across the day

SUMMARY:
Sleep is an essential biological function that impacts nearly every aspect of an athlete's physical and mental health. For athletes, the importance of high-quality sleep cannot be overstated, as it plays a critical role in performance, recovery, and overall well-being. Sleep supports muscle recovery by promoting protein synthesis and the release of growth hormones, essential for healing after intense physical exertion. Furthermore, adequate sleep is crucial for maintaining cognitive sharpness, decision-making abilities, and emotional regulation-all of which are necessary for optimal athletic performance. The study will assess both sleep quality and quantity in baseball players at Columbia University. These tools will help quantify key sleep metrics, including sleep duration, latency (the time it takes to fall asleep), and the number of awakenings during the night. Similarly, the study will analyze dietary patterns using the Automated Self-Administered 24-Hour Dietary Assessment (ASA24), tracking nutrient intake, meal timing, and the consumption of ultra-processed foods. These assessments will establish a baseline from which to measure improvement post-intervention. The intervention will focus on improving diet, time in bed, and light exposure to improve sleep, diet, and performance in collegiate baseball athletes.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate baseball player at Columbia University

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Athletic performance (position-specific for batters and pitchers) | pre and post intervention (4-6 weeks)
  Batters: Baseball radar gun, outcome is exit velocity (speed at which ball leaves the bat, in miles/h) Pitchers: Baseball radar gun measuring velocity (miles/h)
Sleep quality | Nightly for 6 weeks
  Duration (h:min)
Sleep quality | Nightly for 6 weeks
  Sleep stage (%REM, %Deep sleep)
Dietary quality | pre and post intervention (4-6 weeks)
  3-day food recalls (ASA-24)

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) | pre and post intervention (4-6 weeks)
  7 questions, 0-3 points each (not at all to nearly every day); global score 0-21, higher score is worse
Patient Health Questionnaire-9 | pre and post intervention (4-6 weeks)
  9 questions, 0-3 points each (not at all to nearly every day); global score 0-27, higher score is worse
Sport Anxiety Scale-2 | pre and post intervention (4-6 weeks)
  4-point Likert scale (not at all to very much); global score 5-20, higher score is worse
Pitching accuracy | pre and post intervention (4-6 weeks)
  Ratio of strikes to balls (pitchers only)
Isometric wall push | pre and post intervention (4-6 weeks)
  Hand-held dynamometer (pounds) (pitchers only)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Principal Investigator — Columbia University Vagelos College of Physicians & Surgeons
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States